CLINICAL TRIAL: NCT02026453
Title: Pharmacists and Pharmacy Technicians to Improve Admission Medication History Accuracy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Josh Pevnick, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KL2TR000122-00032874; K23AG049181-01 (NIH); KL2TR000122 (NIH)
Record Dates: First submitted 2013-12-31; First posted 2014-01-03 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Adverse Drug Events
Keywords: Adverse drug events
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (No Intervention): Physicians and nurses obtain admission medication history.
- Pharmacist obtains home med hx (Experimental): Pharmacist obtains admission medication history, although usual care practices may also continue.
  Interventions: Other: Pharmacist obtains admission medication history
- Pharm tech obtains home med hx (Experimental): Pharmacy technician obtains admission medication history, although usual care practices may also continue.
  Interventions: Other: Pharmacy technician obtains admission medication history

INTERVENTIONS:
Other: Pharmacist obtains admission medication history
  Arms: Pharmacist obtains home med hx
Other: Pharmacy technician obtains admission medication history
  Arms: Pharm tech obtains home med hx

SUMMARY:
We tested two interventions to improve the accuracy of medication histories obtained at hospital admission. The interventions target elderly and chronically ill patients prone to erroneous medication histories and resultant medication errors. For targeted patients, we tested the effect of using pharmacists and pharmacy technicians to obtain an initial medication history. This was studied using a randomized controlled trial of usual care (which involves nurses and physicians) vs usual care + pharmacists vs usual care + pharmacy technicians to obtain an admission medication history.

The overarching hypothesis was that by leveraging pharmacists and pharmacy technicians we can minimize admission medication history errors and related downstream events.

DETAILED DESCRIPTION:
Importance: Admission medication history (AMH) errors frequently cause medication order errors and patient harm.

Objective: To quantify AMH error reduction achieved when pharmacy staff obtain AMHs before admission medication orders (AMO) are placed.

Design: Three-arm randomized clinical trial. Setting: Large hospital with community and trainee physicians. Population: 306 enrolled patients with complex medical histories. Interventions: In one intervention arm, pharmacists, and in the second intervention arm, pharmacy technicians obtained initial AMHs prior to admission. They obtained and reconciled medication information from multiple sources. All arms, including the control arm, received usual AMH care. This included common process variation occurring in: accuracy of pre-existing medication histories; nurses' ability to obtain AMHs at hospital admission; and admitting physicians' efforts to verify and order from prior AMHs.

Main Outcomes and Measures: The primary outcome was severity-weighted mean AMH error score. To detect AMH errors, all patients received reference standard AMHs, which were compared with intervention and control group AMHs. AMH errors and resultant AMO errors were independently identified and rated by ≥2 investigators as significant, serious or life-threatening. Each error was assigned 1, 4 or 9 points, respectively, to calculate severity-weighted AMH and AMO error scores for each patient.

ELIGIBILITY:
Inclusion criteria:

* Accessed via EHR, were: >=10 chronic prescription medications
* History of acute myocardial infarction or congestive heart failure
* Admission from skilled nursing facility
* History of transplant, or active anticoagulant, insulin, or narrow therapeutic index medications.

Exclusion criteria:(supersedes inclusion criteria)

* Admitted to pediatric, trauma or transplant services with pharmacists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Pevnick, MD, MSHS, Principal Investigator — Cedars-Sinai Health System

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pevnick JM, Palmer KA, Shane R, Wu CN, Bell DS, Diaz F, Cook-Wiens G, Jackevicius CA. Potential benefit of electronic pharmacy claims data to prevent medication history errors and resultant inpatient order errors. J Am Med Inform Assoc. 2016 Sep;23(5):942-50. doi: 10.1093/jamia/ocv171. Epub 2016 Jan 17. PMID 26911817
- [Result] Nguyen CB, Shane R, Bell DS, Cook-Wiens G, Pevnick JM. A Time and Motion Study of Pharmacists and Pharmacy Technicians Obtaining Admission Medication Histories. J Hosp Med. 2017 Mar;12(3):180-183. doi: 10.12788/jhm.2702. PMID 28272596
- [Result] Pevnick JM, Nguyen C, Jackevicius CA, Palmer KA, Shane R, Cook-Wiens G, Rogatko A, Bear M, Rosen O, Seki D, Doyle B, Desai A, Bell DS. Improving admission medication reconciliation with pharmacists or pharmacy technicians in the emergency department: a randomised controlled trial. BMJ Qual Saf. 2018 Jul;27(7):512-520. doi: 10.1136/bmjqs-2017-006761. Epub 2017 Oct 6. PMID 28986515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were medically complex patients admitted to Cedars-Sinai Medical Center, a large university-affiliated hospital, through the emergency department. Enrollment screening occurred Mondays through Thursdays from approximately 11 AM to 8 PM beginning 1/7/2014 through 2/14/2014.
Groups:
- Pharmacist Obtains Home Med hx: Pharmacist obtains admission medication history, although usual care practices may also continue.
  Pharmacist obtains admission medication history
- Pharm Tech Obtains Home Med hx: Pharmacy technician obtains admission medication history, although usual care practices may also continue.
  Pharmacy technician obtains admission medication history
Period: Overall Study
Arm/Group | Usual Care | Pharmacist Obtains Home Med hx | Pharm Tech Obtains Home Med hx
Started | 101 | 103 | 102
Completed | 95 | 94 | 89
Not Completed | 6 | 9 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Pharmacist Obtains Home Med hx | Pharm Tech Obtains Home Med hx | Total
Number analyzed (Participants) | 101 | 103 | 102 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (18) | 72 (16) | 71 (16) | 72 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 54 | 55 | 157
  Male | 53 | 49 | 47 | 149

OUTCOME MEASURES:

1. Primary Outcome: Mean Severity-weighted Admission Medication History (AMH) Error Score
Description: The primary outcome was severity-weighted mean admission medication history (AMH) error score which are weighted error counts. Significant, serious, and life-threatening errors count for 1, 4, and 9 points each, respectively. As such, higher scores indicate either more errors or errors of greater severity. The range includes integers starting with 0 (indicating zero errors) up to infinity. To detect AMH errors, all patients received reference standard AMHs, which were compared with intervention and control group AMHs. AMH errors and resultant AMO errors were independently identified and rated by ≥2 investigators as significant, serious or life-threatening.
Time Frame: Attempted to obtain the day after admission
Measure: Mean (95% Confidence Interval); unit: Mean Severity-weighted AMH Error Score
Arm/Group | Usual Care | Pharmacist Obtains Home Med hx | Pharm Tech Obtains Home Med hx
Number analyzed (Participants) | 95 | 94 | 89
Mean Severity-weighted AMH Error Score | 23 [19.7 to 26.2] | 4.1 [2.7 to 5.5] | 4.1 [2.6 to 5.6]

2. Secondary Outcome: Mean Severity-Weighted Admission Medication Order (AMO) Error Score
Description: The severity-weighted admission medication order (AMO) error score are weighted error counts. Significant, serious, and life-threatening errors count for 1, 4, and 9 points each, respectively. Higher scores indicate either more errors or errors of greater severity. The range includes integers starting with 0 (indicating zero errors) up to infinity. For each AMH error identified, two physicians independently reviewed the relevant medications ordered at hospital admission in the context of the clinical chart. They classified each AMH error as either resulting in no AMO error, or an AMO error of significant, serious, or life-threatening severity. A third physician adjudicated disagreements. In cases where the admitting physician's knowledge of an AMH error was unclear and the orders clinically reasonable, we determined the AMH error did not lead to any AMO error. Because reviewers needed chart access to determine error severity, there was no practicable way to mask study arm.
Time Frame: Attempted to obtain the day after admission
Measure: Mean (95% Confidence Interval); unit: Mean Severity-Weighted AMO Error Score
Arm/Group | Usual Care | Pharmacist Obtains Home Med hx | Pharm Tech Obtains Home Med hx
Number analyzed (Participants) | 95 | 94 | 89
Mean Severity-Weighted AMO Error Score | 6.9 [5.5 to 8.4] | 1.5 [.089 to 2.1] | 1.2 [.067 to 1.7]

ADVERSE EVENTS:
Description: In terms of the Participants at Risk and similar outcomes, please note that "0" signifies that adverse events were not collected or assessed as part of the study. Also, the intervention, which involved having pharmacists and pharmacy technicians talk with patients/families/caregivers and review records in detail, was deemed to represent minimal risk.
Arm/Group | Usual Care | Pharmacist Obtains Home Med hx | Pharm Tech Obtains Home Med hx
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
* Powered on intermediate endpoints
* Only used one site
* Could not practicably mask arm allocation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No